CLINICAL TRIAL: NCT06713291
Title: Prospective, Multicenter, Randomized Controlled Clinical Study of a Novel Sliding Compression Locking Plate in the Treatment of Fresh Femoral Neck Fractures
Brief Title: Clinical Study of a Novel Sliding Compression Locking Plate in the Treatment of Fresh Femoral Neck Fractures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhang Wei, Professor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Chinese PLA General Hosptial
Record Dates: First submitted 2024-11-16; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Fracture of Femoral Neck
Keywords: fracture of neck of femur, sliding compression locking plate, compression screws
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sliding compression locking plate (Experimental): Patients with femoral neck fracture were treated with sliding compression locking plate internal fixation.
  Interventions: Procedure: Sliding compression locking plate
- Three cannulated compression screws (Placebo Comparator): The patients with femoral neck fracture were treated with three cannulated compression screws.
  Interventions: Procedure: Three cannulated compression screws

INTERVENTIONS:
Procedure: Sliding compression locking plate — The patients with femoral neck fracture were treated with three cannulated compression screws or sliding compression locking plate.
  Arms: Sliding compression locking plate
Procedure: Three cannulated compression screws — The patients with femoral neck fracture were treated with three cannulated compression screws.
  Arms: Three cannulated compression screws

SUMMARY:
To verify the safety and efficacy of sliding compression locking plates in the treatment of fresh femoral neck fractures

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 years old, gender is not limited;
2. Patients diagnosed with femoral neck fracture;
3. Patients with indications for internal fixation of femoral neck fracture and able to tolerate surgery;
4. The subject or his legal representative is informed of the nature of the study and agrees to participate in the study.

Exclusion Criteria:

1. Participants who had participated in clinical studies of other drugs, biologics or medical devices before enrollment and did not reach the primary study endpoint time limit;
2. The patient is known to have a history of allergy to one or more implanted materials;
3. Patients determined by researchers to be physically weak or unable to tolerate surgery due to other systemic diseases;
4. Active infection of the hip joint or other parts of the body is determined by the investigator;
5. Diagnosed as metabolic bone disease, radiation bone disease, etc.;
6. Severe hip contracture deformity or severe muscle loss fused to the functional position for a long time without pain;
7. have inflammatory arthritis, such as rheumatoid arthritis, systemic lupus erythematosus arthritis, ankylosing spondylitis, etc.;
8. The patient is mentally incapable or unable to understand the requirements of participating in the study, and it is difficult to cooperate;
9. Other conditions deemed unsuitable for inclusion by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1150 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Femoral neck shortened | 1 year
  The difference in femoral neck length between 1 week post-surgery and 6 months and 12 months post-surgery, measured via X-ray and CT imaging examinations.

SECONDARY OUTCOMES:
Neck shaft angle | 1 year
The effectiveness of guide pin implantation | 1 day
  For the cohort treated with three cannulated compression screws, the effectiveness of guide pin implantation is categorized into three parallel, two parallel, and non-parallel arrangements，which will be measured during the surgery.
Time of operation | 1 day
Blood loss | 1 day
Bone union | 1 year
Zarit Burden Interview（ZBI） | 1 year
  The Zarit Burden Interview (ZBI) is a commonly used assessment tool designed to quantify the psychological and emotional burden experienced by caregivers who provide care for individuals with cognitive or functional impairments. Developed by Zarit and colleagues, the scale consists of 22 items that cover various aspects of caregiver burden, such as time pressure, emotional strain, and social isolation. The scoring ranges from 0 to 88, with higher scores indicating a greater level of caregiving burden. This tool aids healthcare professionals in identifying the psychological stress faced by caregivers and provides appropriate support and interventions to improve their mental health and quality of life.
SF-36 Score | 1 year
  The SF-36 (Short Form 36 Health Survey) is a widely used generic health status assessment tool developed by the Medical Outcomes Study (MOS) Group. The scale is designed to comprehensively evaluate health-related quality of life, encompassing eight dimensions: physical functioning, social functioning, role limitations due to physical health, role limitations due to emotional problems, bodily pain, mental health, vitality, and general health perceptions. Each dimension consists of several items, and scores are derived by summing the scores of these items, typically converted to a 0 to 100 percent scale, with 100 representing the best possible health state. These eight dimension scores can be combined to form two summary scores: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hosptial, Beijing, China

IPD SHARING:
Plan to Share IPD: No